CLINICAL TRIAL: NCT04120636
Title: Phase I Study of Sequestered Transscleral, Controlled-Release Celecoxib Delivered Via Episcleral Reservoir for Treatment of Macular Edema & Inflammatory Disorders of the Eye Posterior Pole Including Sclera, Choroid, Retina or Vitreous
Brief Title: Phase I Study of Episcleral Celecoxib for Treatment of Macular Edema and Inflammatory Disorders of the Posterior Pole
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targeted Therapy Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3TCEL-02
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Macula Edema; Radiation Retinopathy; Branch Retinal Vein Occlusion; Epiretinal Membrane; Central Serous Retinopathy With Pit of Optic Disc; Commotio Retinae; Vitritis
Keywords: Macula Edema; Radiation Retinopathy; Branch Retinal Vein Occlusion; Epiretinal Membrane; Central Serous Retinopathy with Pit of Optic Disc; Commotio Retinae; Vitritis
MeSH Terms: conditions — Retinal Vein Occlusion; Epiretinal Membrane; Uveitis, Intermediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I open label study (Experimental): Drug: Episcleral Celecoxib
  Other Names:
  * Sequestered, Transscleral, Controlled-Release Celecoxib
  * Sustained Release Transscleral Celecoxib
  Interventions: Drug: Episcleral Celecoxib

INTERVENTIONS:
Drug: Episcleral Celecoxib — Sustained Release Transscleral Celecoxib
  Other Names: Sustained Release Transscleral Celecoxib

SUMMARY:
This phase I trial will assess primarily the safety and secondarily the anti-inflammatory and anti-neovascular effect of Episcleral Celecoxib in patients suffering from macular edema and other inflammatory disorders of the retina, choroid and vitreous.

DETAILED DESCRIPTION:
This phase I trial will assess primarily the safety and secondarily anti-inflammatory/neovascular effect of Episcleral Celecoxib in patients suffering from macular edema & inflammatory disorders of the eye posterior pole Including sclera, choroid, retina, or vitreous. Celecoxib is a specific cyclooxygenase-2 inhibitor that possesses anti-angiogenic, anti-inflammatory, and anti-fibrotic properties. Non-clinical studies have documented the activity of Celecoxib in reducing leakage of the blood-retina barrier as well as inhibiting vascular endothelial growth factor (VEGF) and prostaglandin E2 (PGE2) expression in the retina of diabetic rats. The underlying mechanisms for its anti-inflammatory and anti-angiogenic properties have been extensively characterized. The investigators hypothesize that Episcleral Celecoxib is safe, tolerable and that its anti-inflammatory/anti-neovascular activity will reduce macular edema and improve vision in patients with macular edema. Objective: to primarily assess the safety, tolerability and pharmacokinetics of Episcleral Celecoxib in patients with macular edema and other inflammatory disorders of the posterior pole including retina, choroid and vitreous to secondarily assess efficacy in reducing macular edema and improving visual function. Methods: The main outcome of the study is safety assessment. Secondary outcomes are assessment of visual acuity and anatomical changes in the macula as measured via optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Visual acuity letter score in study eye < 70 and ≥ 25 letters (approximate Snellen equivalent 20/32 to 20/320);
* Ophthalmoscopic evidence of center-involved macular edema, within the central subfield (CSF); • Inflammatory disorders of the sclera, choroid, retina or vitreous

Exclusion Criteria:

* Inability to understand informed consent, cooperate with testing or return to follow up visits;
* Pregnant or lactating women;
* Co-existent ocular disorder of the cornea, lens or media that will interfere with assessment of safety or efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of the study is ocular safety assessment as measured by comprehensive ophthalmic exam. | 12 Months
  The primary outcome measure of the study is ocular safety assessment as measured by comprehensive ophthalmic exam.

SECONDARY OUTCOMES:
A secondary outcome is assessment of visual acuity. | 12 Months
  A secondary outcome is assessment of visual acuity.
A secondary outcome is assessment of anatomical changes in the macula as measured via optical coherence tomography (OCT). | 12 Months
  A secondary outcome is assessment of anatomical changes in the macula as measured via optical coherence tomography (OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Leng, MD, Principal Investigator — Stanford Medicine Ophthalmology [Recruiting]
Locations (1):
- Stanford Medicine Ophthalmology, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No